CLINICAL TRIAL: NCT02154191
Title: Level of Activity in Lumbar Spinal Stenosis Patients Pre- and Post-surgery: a Non-randomized Controlled Before-after Trial
Brief Title: Level of Activity in Lumbar Spinal Stenosis Patients Pre- and Post-surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: University of Manitoba (Other)
Collaborators: Gibson Orthopaedic Fund for Research and Education (Other)
Responsible Party: Principal Investigator, Dr. Steven Passmore, Steven Passmore, DC, PhD, University of Manitoba
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: H2014:176
Record Dates: First submitted 2014-05-23; First posted 2014-06-03 (Estimated); Last update posted 2015-06-08 (Estimated); Status verified 2015-06

CONDITIONS: Spinal Stenosis
Keywords: Lumbosacral Region; Sedentary Lifestyle; Surgical Procedure, Operative
MeSH Terms: conditions — Spinal Stenosis; Sedentary Behavior | interventions — Surgical Procedures, Operative

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Surgical Intervention Group (Experimental): The Surgical Intervention Group will undergo the routine surgical procedures taken for patients requiring surgery for degenerative lumbar spinal stenosis.
  Interventions: Procedure: Surgical Intervention
- Non-Intervention Group (Control) (No Intervention): No Intervention.This group will consist of patients wait listed for surgery but further back in the queue.

INTERVENTIONS:
Procedure: Surgical Intervention — The clinical intervention in this study is the routine surgical procedures taken for patients requiring surgery for degenerative lumbar spinal stenosis.
  Arms: Surgical Intervention Group

SUMMARY:
The purpose of the proposed research is to explore the relationship between objectively measured physical activity and surgical intervention for lumbar spinal stenosis (LSS). Our primary hypothesis is that post-surgery, LSS patients will demonstrate increased physical activity compared to their baseline assessment. A non-intervention control group will be measured at the same time intervals as the surgical group to look at test re-test reliability. In the event that our hypothesis is rejected, and surgery does not lead to a decrease in sedentary behaviour analysis of questionnaire-based sedentary behaviour measures and objective activity-based measurement can examine the relationship between self-report and actual performance-based objective measures. The primary objective of our proposal is to determine if surgical intervention leads to increased activity, and decreased sedentary behaviour. The findings of the proposed research will inform healthcare stakeholders that if surgery alone does not lead to increased activity, a more concerted research effort may need to be made for post-surgical rehabilitation, lifestyle and physical activity counselling so that post-surgical patients may make changes toward leading more active and productive lives.

DETAILED DESCRIPTION:
Apparatus:

Activity Monitors: The ActiGraph GT3X+ monitor (ActiGraph, Pensacola, FL) has been shown to be reliable and to have good validity under both laboratory and free living conditions. It is one of the most widely respected monitors used for measuring physical activity and sedentary behaviour and is currently being used in an intervention trial with patients with LSS . The GT3X+ monitor includes a triaxial accelerometer, an inclinometer and light sensor. It is capable of measuring activity counts, steps, position relative to gravity and can discriminate between day and night. This accelerometer based sensor system does not impede normal movement and can be worn throughout the day on the waistband, in virtually all environments, except in water. The wGT3X+ activity monitor has the capacity to collect data at up to 100Hz.

Procedure:

Each participant will be given an ActiGraph wGT3X+ activity monitor with instructions to wear the monitor during waking hours over 7 consecutive days except when bathing, showering or swimming. Each ActiGraph monitor will be fastened to a belt over the anterior axillary line at the right hip as per the manufacturer's recommendations and initialized to collect data in 1s epochs. They will also be asked to complete log sheets recording the time they put the monitor on and take it off each day. Participants will complete 2 separate 7-day bouts, six weeks apart.

For the surgical group the ActiGraph will be used in the week leading up to their surgical intervention. The follow-up will occur 6-weeks post surgery. For the no intervention group the ActiGraph will be used in the week immediately after it is determined they are a surgical candidate, and the follow-up will occur 6-weeks later while they are on the surgical waitlist.

Pre-Surgery test:

They will receive the device at a pre-surgical assessment when they will complete their baseline questionnaires, and they will return the device upon their presentation for scheduled surgery.

Post-Surgery test:

When the patient presents for their 6-week post surgical follow-up they will again receive the device, complete questionnaire forms, and be given the device with a postage-paid Express Post envelope to return the monitor to the researchers once they are done with it. Upon arrival of the device, the participant compensation will be issued.

Pre-No Intervention test:

Immediately following the assessment visit when it is determined that the patient is a surgical candidate they will receive the device and complete their baseline questionnaires. In addition, patients will be given a postage-paid Express Post envelope to return the monitor to the researchers once they are done with the it.

Post-No Intervention test:

Six weeks later, the patient will be asked to report to the laboratory where they will again receive the device, complete questionnaire forms, and be given the device with a postage-paid Express Post envelope to return the monitor to the researchers once they are done with it. Upon arrival of the device, the participant compensation will be issued.

Statistical Analysis:

To identify possible explanatory variables, multiple regression will be used to determine relationships between physical activity and sedentary behaviour data (e.g., number of minutes of sedentary, light, moderate physical activity/day, maximum number of consecutive minutes at or above 100 activity counts/ min, maximum sedentary bout length) with demographic factors such as age, duration of diagnosis, body mass index, pain ratings.

Separate paired student's t-tests will be used to compare participants to themselves in terms baseline and follow-up questionnaire scores. Separate unpaired student's t-tests will compare questionnaire based outcome measure scores between groups pre and post intervention. Repeated measures analysis of variance will be used to compare pre- and post-intervention measurements of physical activity and sedentary behaviour within and between groups. Specifically, for all ActiGraph recorded measures separate 2 Group (Surgery, NI) x 2 Time (pre, post) analysis of variance (ANOVA) designs will be employed. Post-hoc analysis will be performed on effects involving more than two means, as needed, using Tukey's Honestly Significant Difference (HSD).

To compare the agreement between the self-report measures and the direct activity monitor data, intra-class correlation (ICC) two-way mixed models will be used.

Adverse Events/Serious Adverse Events:

While this study includes clinical intervention the outcome measures of interest pre- and post-surgery would not be predicted to yield any adverse events. The surgical procedures used are not considered part of the experimental design. The clinical intervention in this study is the routine surgical procedures taken for patients requiring surgery for degenerative lumbar spinal stenosis. If the patients were not enrolled in the study they would be under equal risk for adverse events as a result of the clinical intervention.

Planned Dissemination:

The results of this study will be prepared for dissemination first at relevant clinical and scientific conferences. Subsequently, this work will be submitted to a peer-reviewed journal for consideration of publication.

Additional Ethical Aspects of Protocol:

Potential Benefits to Participants and Others:

The potential benefits of participation to participants include receiving $10 parking reimbursement, on two occasions, and an online gift card for $40 from a grocery store. There are no other direct benefits for participating in this study.

Indirect benefits include knowledge that they have contributed to the advancement of scientific understanding the relationship of physical activity pre and post-surgical intervention.

There are no direct benefits to others. Indirect benefits include those to the scientific community through the planned dissemination of the work. The results of this study will be prepared for dissemination first at relevant clinical and scientific conferences. Subsequently, this work will be submitted to a peer reviewed journal for consideration of publication.

Potential harms to Participants and Others:

There is no anticipated potential harm for participants in regard to outcome measure completion. In regard to surgical intervention the risks and potential harms are equal to those of the patient having surgery outside the research study. All patients recruited for this study would otherwise receive the surgery even if not enrolled in the study.

To protect participant privacy all data collected will be coded and put into database format. All data will be de-identified and kept on a single study computer at each site which is password protected and located in a locked office. As such, access to study subject information/data will be highly safeguarded and can only be accessed by Dr. Passmore. Any paper forms and questionnaires will be kept in a locked cabinet in a locked room. Identifying information that will be collected is the subject's name, contact information and date of birth.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed clinical diagnosis of lumbar spinal stenosis through diagnostic imaging and clinical testing/history from a spine surgeon
* Considered pre-surgical but in need of surgery (surgical necessity also confirmed by a spine surgeon)

Exclusion Criteria:

* Not in immediate surgical need
* No diagnosis of degenerative lumbar spinal stenosis.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2014-06; Primary Completion 2016-06 (Estimated)

PRIMARY OUTCOMES:
Activity Measure - Volume | Change from Baseline Activity Measures at 6 weeks (post-surgery or post non-intervention)
  Daily physical activity data collected by the ActiGraph wGT3X+ activity monitor will be analyzed and described using volume (e.g., activity counts/day).
Activity Measure - Rate | Change from Baseline Activity Measures at 6 weeks (post-surgery or post non-intervention)
  Daily physical activity data collected by the ActiGraph wGT3X+ activity monitor will be analyzed and described using rate (e.g., average steps/minute/day).
Activity Measure - Time Indicators | Change from Baseline Activity Measures at 6 weeks (post-surgery or post non-intervention)
  Daily physical activity data collected by the ActiGraph wGT3X+ activity monitor will be analyzed and described using time indicators (e.g., time spent in sedentary, light, moderate and high intensity physical activity categories/day) using standard cut-point thresholds.
Activity Measure - Maximum Continuous Daily Activity | Change from Baseline Activity Measures at 6 weeks (post-surgery or post non-intervention)
  The maximum number of consecutive minutes at or above 100 activity counts/min (a threshold thought to represent low intensity activity) with no more than 1 min of activity below this low intensity threshold will be determined along with the average duration of activity bouts/day.
Activity Measure - Sedentary Bout Length | Change from Baseline Activity Measures at 6 weeks (post-surgery or post non-intervention)
  Collected by ActiGraph wGT3X+ activity monitor
Activity Measure - Maximum Bout Length | Change from Baseline Activity Measures at 6 weeks (post-surgery or post non-intervention)
  Collected by ActiGraph wGT3X+ activity monitor
Self-Report Measures - Swiss Spinal Stenosis Scale | Change between responses collected at baseline, and 6 weeks later for both groups.
  Questionnaire based outcome measures will be used to subjectively quantify baseline differences between all participants in the Surgery or NI groups.
Self-Report Measures - Quadruple Numeric Rating Scale (QNRS) | Change between responses collected at baseline, and 6 weeks later for both groups.
  Questionnaire based outcome measures will be used to subjectively quantify baseline differences between all participants in the Surgery or NI groups.
Self-Report Measures - Fear Avoidance Belief Questionnaire (FABQ) | Change between responses collected at baseline, and 6 weeks later for both groups.
  Questionnaire based outcome measures will be used to subjectively quantify baseline differences between all participants in the Surgery or NI groups.
Self-Report Measures - Sedentary Behaviors Questionnaire (SBQ) | Change between responses collected at baseline, and 6 weeks later for both groups.
  Questionnaire based outcome measures will be used to subjectively quantify baseline differences between all participants in the Surgery or NI groups.
Self-Report Measures - Short Form Health Survey (SF-36) | Change between responses collected at baseline, and 6 weeks later for both groups.
  Questionnaire based outcome measures will be used to subjectively quantify baseline differences between all participants in the Surgery or NI groups.

CONTACTS AND LOCATIONS:
Overall Officials: Steven Passmore, DC, PhD, Principal Investigator — University of Manitoba
Locations (1):
- Health Sciences Centre (Rehab Hospital, RR-309), Winnipeg, Manitoba, Canada

REFERENCES:
- [Background] Aadland E, Andersen JR, Anderssen SA, Kvalheim OM. Physical activity versus sedentary behavior: associations with lipoprotein particle subclass concentrations in healthy adults. PLoS One. 2013 Dec 27;8(12):e85223. doi: 10.1371/journal.pone.0085223. eCollection 2013. PMID 24386464
- [Background] Brown HE, Ryde GC, Gilson ND, Burton NW, Brown WJ. Objectively measured sedentary behavior and physical activity in office employees: relationships with presenteeism. J Occup Environ Med. 2013 Aug;55(8):945-53. doi: 10.1097/JOM.0b013e31829178bf. PMID 23887700
- [Background] Ciol MA, Deyo RA, Howell E, Kreif S. An assessment of surgery for spinal stenosis: time trends, geographic variations, complications, and reoperations. J Am Geriatr Soc. 1996 Mar;44(3):285-90. doi: 10.1111/j.1532-5415.1996.tb00915.x. PMID 8600197
- [Background] Conway J, Tomkins CC, Haig AJ. Walking assessment in people with lumbar spinal stenosis: capacity, performance, and self-report measures. Spine J. 2011 Sep;11(9):816-23. doi: 10.1016/j.spinee.2010.10.019. Epub 2010 Dec 8. PMID 21145292
- [Background] Haskell WL, Lee IM, Pate RR, Powell KE, Blair SN, Franklin BA, Macera CA, Heath GW, Thompson PD, Bauman A. Physical activity and public health: updated recommendation for adults from the American College of Sports Medicine and the American Heart Association. Med Sci Sports Exerc. 2007 Aug;39(8):1423-34. doi: 10.1249/mss.0b013e3180616b27. PMID 17762377
- [Background] Jenis LG, An HS. Spine update. Lumbar foraminal stenosis. Spine (Phila Pa 1976). 2000 Feb 1;25(3):389-94. doi: 10.1097/00007632-200002010-00022. PMID 10703115
- [Background] Katz JN, Harris MB. Clinical practice. Lumbar spinal stenosis. N Engl J Med. 2008 Feb 21;358(8):818-25. doi: 10.1056/NEJMcp0708097. No abstract available. PMID 18287604
- [Background] Otani K, Takegami M, Fukumori N, Sekiguchi M, Onishi Y, Yamazaki S, Ono R, Otoshi K, Hayashino Y, Fukuhara S, Kikuchi S, Konno S; LOHAS Research Group. Locomotor dysfunction and risk of cardiovascular disease, quality of life, and medical costs: design of the Locomotive Syndrome and Health Outcome in Aizu Cohort Study (LOHAS) and baseline characteristics of the study population. J Orthop Sci. 2012 May;17(3):261-71. doi: 10.1007/s00776-012-0200-5. Epub 2012 Apr 12. PMID 22526710
- [Background] Pratt RK, Fairbank JC, Virr A. The reliability of the Shuttle Walking Test, the Swiss Spinal Stenosis Questionnaire, the Oxford Spinal Stenosis Score, and the Oswestry Disability Index in the assessment of patients with lumbar spinal stenosis. Spine (Phila Pa 1976). 2002 Jan 1;27(1):84-91. doi: 10.1097/00007632-200201010-00020. PMID 11805642
- [Background] Pryce R, Johnson M, Goytan M, Passmore S, Berrington N, Kriellaars D. Relationship between ambulatory performance and self-rated disability in patients with lumbar spinal stenosis. Spine (Phila Pa 1976). 2012 Jul 1;37(15):1316-23. doi: 10.1097/BRS.0b013e31824a8314. PMID 22261635
- [Background] Rabinovich RA, Louvaris Z, Raste Y, Langer D, Van Remoortel H, Giavedoni S, Burtin C, Regueiro EM, Vogiatzis I, Hopkinson NS, Polkey MI, Wilson FJ, Macnee W, Westerterp KR, Troosters T; PROactive Consortium. Validity of physical activity monitors during daily life in patients with COPD. Eur Respir J. 2013 Nov;42(5):1205-15. doi: 10.1183/09031936.00134312. Epub 2013 Feb 8. PMID 23397303
- [Background] Santos-Lozano A, Marin PJ, Torres-Luque G, Ruiz JR, Lucia A, Garatachea N. Technical variability of the GT3X accelerometer. Med Eng Phys. 2012 Jul;34(6):787-90. doi: 10.1016/j.medengphy.2012.02.005. Epub 2012 Mar 13. PMID 22417978
- [Background] Schulte TL, Schubert T, Winter C, Brandes M, Hackenberg L, Wassmann H, Liem D, Rosenbaum D, Bullmann V. Step activity monitoring in lumbar stenosis patients undergoing decompressive surgery. Eur Spine J. 2010 Nov;19(11):1855-64. doi: 10.1007/s00586-010-1324-y. Epub 2010 Feb 26. PMID 20186442
- [Background] Stucki G, Daltroy L, Liang MH, Lipson SJ, Fossel AH, Katz JN. Measurement properties of a self-administered outcome measure in lumbar spinal stenosis. Spine (Phila Pa 1976). 1996 Apr 1;21(7):796-803. doi: 10.1097/00007632-199604010-00004. PMID 8779009
- [Background] Tomkins-Lane CC, Conway J, Hepler C, Haig AJ. Changes in objectively measured physical activity (performance) after epidural steroid injection for lumbar spinal stenosis. Arch Phys Med Rehabil. 2012 Nov;93(11):2008-14. doi: 10.1016/j.apmr.2012.05.014. Epub 2012 May 31. PMID 22659537
- [Background] Tomkins-Lane CC, Haig AJ. A review of activity monitors as a new technology for objectifying function in lumbar spinal stenosis. J Back Musculoskelet Rehabil. 2012;25(3):177-85. doi: 10.3233/BMR-2012-0325. PMID 22935856
- [Background] Tomkins-Lane CC, Lafave LM, Parnell JA, Krishnamurthy A, Rempel J, Macedo LG, Moriartey S, Stuber KJ, Wilson PM, Hu R, Andreas YM. The spinal stenosis pedometer and nutrition lifestyle intervention (SSPANLI) randomized controlled trial protocol. BMC Musculoskelet Disord. 2013 Nov 14;14:322. doi: 10.1186/1471-2474-14-322. PMID 24228747
- [Background] Troiano RP, Berrigan D, Dodd KW, Masse LC, Tilert T, McDowell M. Physical activity in the United States measured by accelerometer. Med Sci Sports Exerc. 2008 Jan;40(1):181-8. doi: 10.1249/mss.0b013e31815a51b3. PMID 18091006
- [Background] Tudor-Locke C, Brashear MM, Johnson WD, Katzmarzyk PT. Accelerometer profiles of physical activity and inactivity in normal weight, overweight, and obese U.S. men and women. Int J Behav Nutr Phys Act. 2010 Aug 3;7:60. doi: 10.1186/1479-5868-7-60. PMID 20682057
- [Background] Van Remoortel H, Raste Y, Louvaris Z, Giavedoni S, Burtin C, Langer D, Wilson F, Rabinovich R, Vogiatzis I, Hopkinson NS, Troosters T; PROactive consortium. Validity of six activity monitors in chronic obstructive pulmonary disease: a comparison with indirect calorimetry. PLoS One. 2012;7(6):e39198. doi: 10.1371/journal.pone.0039198. Epub 2012 Jun 20. PMID 22745715
- [Background] Warburton DE, Nicol CW, Bredin SS. Health benefits of physical activity: the evidence. CMAJ. 2006 Mar 14;174(6):801-9. doi: 10.1503/cmaj.051351. PMID 16534088
- [Background] Wetten AA, Batterham M, Tan SY, Tapsell L. Relative validity of 3 accelerometer models for estimating energy expenditure during light activity. J Phys Act Health. 2014 Mar;11(3):638-47. doi: 10.1123/jpah.2011-0167. Epub 2013 Feb 8. PMID 23417054
- [Background] Winter CC, Brandes M, Muller C, Schubert T, Ringling M, Hillmann A, Rosenbaum D, Schulte TL. Walking ability during daily life in patients with osteoarthritis of the knee or the hip and lumbar spinal stenosis: a cross sectional study. BMC Musculoskelet Disord. 2010 Oct 12;11:233. doi: 10.1186/1471-2474-11-233. PMID 20939866
- [Background] World Health Organization. Towards a Common Language for Functioning, Disability and Health. 2002